CLINICAL TRIAL: NCT05333107
Title: A Study Investigating the Pharmacokinetic Properties When Dosing Different Formulations of NNC0385-0434 to Healthy Male Participants - Oral Formulation II
Brief Title: A Research Study Looking at New Protein-based Tablets in Healthy Men - Oral Formulation II
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9501-4869; U1111-1271-3953 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteers; High Cholesterol
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Participants will receive oral dose of NNC0385-0434 G tablet for the initial 10-day treatment period (period 1) and the NNC0385-0434 B tablet orally in the 5-day treatment period (period 2).
  Interventions: Drug: NNC0385-0434 G; Drug: NNC0385-0434 B
- Sequence 2 (Experimental): Participants will receive oral dose of NNC0385-0434 G tablet for the initial 10-day treatment period (period 1) and the NNC0385-0434 F tablet orally in the 5-day treatment period (period 2).
  Interventions: Drug: NNC0385-0434 G; Drug: NNC0385-0434 F
- Sequence 3 (Experimental): Participants will receive oral dose of NNC0385-0434 F tablet for the initial 10-day treatment period (period 1) and the NNC0385-0434 B tablet orally in the 5-day treatment period (period 2).
  Interventions: Drug: NNC0385-0434 F; Drug: NNC0385-0434 B
- Sequence 4 (Experimental): Participants will receive oral dose of NNC0385-0434 F tablet for the initial 10-day treatment period (period 1) and the NNC0385-0434 G tablet orally in the 5-day treatment period (period 2).
  Interventions: Drug: NNC0385-0434 G; Drug: NNC0385-0434 F
- Sequence 5 (Experimental): Participants will receive oral dose of NNC0385-0434 B tablet for the initial 10-day treatment period (period 1) and the NNC0385-0434 G tablet orally in the 5-day treatment period (period 2).
  Interventions: Drug: NNC0385-0434 G; Drug: NNC0385-0434 B
- Sequence 6 (Experimental): Participants will receive oral dose of NNC0385-0434 B tablet for the initial 10-day treatment period (period 1) and the NNC0385-0434 F tablet orally in the 5-day treatment period (period 2).
  Interventions: Drug: NNC0385-0434 F; Drug: NNC0385-0434 B

INTERVENTIONS:
Drug: NNC0385-0434 G — Participants will receive oral dose of NNC0385-0434 G tablet either for the initial 10-day treatment period (period 1) or 5-day treatment period (period 2).
  Arms: Sequence 1; Sequence 2; Sequence 4; Sequence 5
Drug: NNC0385-0434 F — Participants will receive oral dose of NNC0385-0434 F tablet either for the initial 10-day treatment period (period 1) or 5-day treatment period (period 2).
  Arms: Sequence 2; Sequence 3; Sequence 4; Sequence 6
Drug: NNC0385-0434 B — Participants will receive oral dose of NNC0385-0434 B tablet either for the initial 10-day treatment period (period 1) or 5-day treatment period (period 2).
  Arms: Sequence 1; Sequence 3; Sequence 5; Sequence 6

SUMMARY:
In this study, the study drug 'NNC0385-0434' will be tested in 3 different tablet formulations. These formulations are being tested for the treatment of hypercholesterolemia (high cholesterol). Participants will only receive 2 of the 3 tablet formulations. The treatments participants get are decided by chance. Participants will receive 1 formulation for 10 days (first treatment period) and the other formulation for 5 days (second treatment period). The study will last up to 96 days. Only men can participate in this clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 18-64 years (both inclusive) at the time of signing informed consent
* Body mass index between 20.0 and 32.0 kilogram per meter square (both inclusive)
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Known or suspected hypersensitivity to study interventions or related products
* Use of prescription medicinal products or non-prescription drugs (including herbal products and vaccines), except routine vitamins and topical medications not reaching the systemic circulation, within 14 days prior to the day of screening
* Any disorder which in the investigator's opinion might jeopardise participant safety or compliance with the protocol
* Presence of clinically significant gastrointestinal disorders potentially affecting absorption of drugs and/or nutrients, as judged by the investigator
* History of major surgical procedures involving the stomach potentially affecting absorption of study products (example: subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery)

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
AUC0-24h,NNC0385-0434,day10; area under the plasma concentrationtime curve during a dosing interval | From 0 to 24 hours after dose administration on visit 2, day 10
  Measured in h * nmol/L

SECONDARY OUTCOMES:
Cmax,NNC0385-0434,day10; maximum observed plasma concentration of NNC0385-0434 | From 0 to 24 hours after dose administration on visit 2, day 10
  Measured in nmol/L
tmax,NNC0385-0434,day10; time from dose administration to maximum observed plasma concentration of NNC0385- 0434 | From 0 to 24 hours after dose administration on visit 2, day 10
  Measured in hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (2):
- United States (2):
  - Altasciences, Cypress, California
  - Altasciences Clinical Los Angeles, Inc., Los Angeles, California

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com